CLINICAL TRIAL: NCT01287403
Title: Response of Alkylresorcinols and Other Biomarkers to Different Cereals
Brief Title: Response of Alkylresorcinols to Different Cereals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, CDUuser, MD, PhD, Société des Produits Nestlé (SPN)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 10.14 MET
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Cereals; Alkylresorcinols; Betaine; Phenolics; Plasma and urine cereal phytochemicals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Refined wheat flour (Placebo Comparator): A negative control flour to serve as a reference.
  Interventions: Other: Esterase wholegrain wheat flour; Other: Wholegrain wheat flour; Other: Liquid whole grain wheat flour; Other: Wholegrain barley flour; Other: Liquid wholegrain barley flour
- Esterase wholegrain wheat flour (Active Comparator): Wholegrain wheat flour treated with esterases to release phenolics (positive control for phenolic acids)
  Interventions: Other: Refined wheat flour; Other: Wholegrain wheat flour; Other: Liquid whole grain wheat flour; Other: Wholegrain barley flour; Other: Liquid wholegrain barley flour
- Wholegrain wheat flour (Experimental): Flour with unknown response
  Interventions: Other: Refined wheat flour; Other: Esterase wholegrain wheat flour; Other: Liquid whole grain wheat flour; Other: Wholegrain barley flour; Other: Liquid wholegrain barley flour
- Liquid whole grain wheat flour (Experimental): Test flour with unknown response.
  Interventions: Other: Refined wheat flour; Other: Esterase wholegrain wheat flour; Other: Wholegrain wheat flour; Other: Wholegrain barley flour; Other: Liquid wholegrain barley flour
- Wholegrain barley flour (Experimental): Test flour with unknown response.
  Interventions: Other: Refined wheat flour; Other: Esterase wholegrain wheat flour; Other: Wholegrain wheat flour; Other: Liquid whole grain wheat flour; Other: Liquid wholegrain barley flour
- Liquid wholegrain barley flour (Experimental): Test flour with unknown response.
  Interventions: Other: Refined wheat flour; Other: Esterase wholegrain wheat flour; Other: Wholegrain wheat flour; Other: Liquid whole grain wheat flour; Other: Wholegrain barley flour

INTERVENTIONS:
Other: Refined wheat flour — A treated cereal flour mixed with milk.
  Arms: Esterase wholegrain wheat flour; Liquid whole grain wheat flour; Liquid wholegrain barley flour; Wholegrain barley flour; Wholegrain wheat flour
Other: Esterase wholegrain wheat flour — A treated cereal flour mixed with milk.
  Arms: Liquid whole grain wheat flour; Liquid wholegrain barley flour; Refined wheat flour; Wholegrain barley flour; Wholegrain wheat flour
Other: Wholegrain wheat flour — A treated cereal flour mixed with milk.
  Arms: Esterase wholegrain wheat flour; Liquid whole grain wheat flour; Liquid wholegrain barley flour; Refined wheat flour; Wholegrain barley flour
Other: Liquid whole grain wheat flour — A treated cereal flour mixed with milk.
  Arms: Esterase wholegrain wheat flour; Liquid wholegrain barley flour; Refined wheat flour; Wholegrain barley flour; Wholegrain wheat flour
Other: Wholegrain barley flour — A treated cereal flour mixed with milk.
  Arms: Esterase wholegrain wheat flour; Liquid whole grain wheat flour; Liquid wholegrain barley flour; Refined wheat flour; Wholegrain wheat flour
Other: Liquid wholegrain barley flour — A treated cereal flour mixed with milk.
  Arms: Esterase wholegrain wheat flour; Liquid whole grain wheat flour; Refined wheat flour; Wholegrain barley flour; Wholegrain wheat flour

SUMMARY:
Cereal grains contain a wide variety of different phytochemicals which may play different roles in physiology. Their response in plasma and urine after a meal is poorly defined for most cereals. This study will investigate the plasma response and urinary excretion of cereal compounds after eating 6 different types of cereal preparation, with a focus on alkylresorcinols.

DETAILED DESCRIPTION:
This was a cross-over, randomized, double blind study with 6 arms (flours of different composition). Thirteen subjects completed the trial, where 100 g of each flour, mixed with 300 mL milk, was fed to all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal-overweight (BMI 19-28 kg/m2)
* Non-smokers

Exclusion Criteria:

* Regular consumers of wholegrain cereals
* Allergy to cereal or milk products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair B Ross, PhD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- NESTEC / Clinical Development Unit / Metabolic Unit, Lausanne, Canton of Vaud, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 healthy subjects were recruited within the staff of the Nestle Research Center. After being informed, by written and orally, on the aims, methods, risk/benefit ratio for the study, they signed an informed consent form and underwent a medical visit screening as per protocol
Pre-assignment Details: Thirteen subjects completed the trial, where 100 g of each flour, mixed with 300 mL milk, was fed to all subjects.
  Subjects avoided foods containing whole grains for one week prior, and 36 h before the start of each treatment, to avoid all phenolic-rich foods (e.g. coffee, tea, chocolate, most fruits and vegetables).
Groups:
- Six Products (Flours) Assigned Randomly (Cross Over): In a crossover design, all subjects were administered the 6 following products in a randomized order:
  Esterase wholegrain wheat flour: a cereal flour treated with esterases to release phenolics (positive control for phenolic acids).
  Refined wheat flour: a treated cereal flour mixed with milk (negative control).
  Liquid whole grain wheat flour: a treated cereal flour mixed with milk.
  Liquid wholegrain barley flour: a treated cereal flour mixed with milk.
  Wholegrain wheat flour: a treated cereal flour mixed with milk.
  Wholegrain barley flour: a treated cereal flour mixed with milk.
Period: Diet Restriction (7 Days)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 14
Completed | 14
Not Completed | 0
Period: 1st Intervention (1 Day)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 14
Completed | 13 (The adverse event was linked to the intake of "refined wheat flour")
Not Completed | 1
Not completed — Adverse Event | 1
Period: Washout 7 Days
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: 2nd Intervention (1 Day)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: 3rd Intervention (1 Day)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: 4th Intervention (1 Day)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: 5th Intervention (1 Day)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0
Period: 6th and Last Intervention (1 Day)
Arm/Group | Six Products (Flours) Assigned Randomly (Cross Over)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects were recruited within the staff of the Nestlé Research Center between February and June 2011.
Groups:
- Entire Study Population: Includes groups randomized to receive either esterase wholegrain wheat flour first or liquid wholegrain wheat flour first or liquid wholegrain barley flour first or refined wheat flour first or wholegrain wheat flour first or wholegrain barley flour first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age, Customized [Number; unit: participants]
  < 18 years | 0
  between 18 and 55 years | 14
  > 55 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  Switzerland | 14

OUTCOME MEASURES:

1. Primary Outcome: Plasma Alkylresorcinol Compounds
Description: Area under the curve (AUC) over baseline of alkylresorcinol compounds are measured for the 6 interventional arms. Time points are: t = 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24 and 48 h after product intake.
Time Frame: From 0 to 48 h post dose.
Measure: Mean (Standard Deviation); unit: nmol/L*h
Groups:
- Esterase Whole Grain Wheat Flour: A cereal flour treated with esterase to release phenolics (positive control for phenolic acids).
- Refined Wheat Flour: A treated cereal flour mixed with milk(negative control).
Arm/Group | Esterase Whole Grain Wheat Flour | Refined Wheat Flour | Liquid Whole Grain Wheat Flour | Liquid Wholegrain Barley Flour | Wholegrain Wheat Flour | Wholegrain Barley Flour
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13 | 13
nmol/L*h | 19357 (7509) | 1548 (698) | 17307 (5914) | 5385 (2642) | 17139 (6386) | 5634 (2478)

2. Secondary Outcome: Plasma and Urinary Betaine
Time Frame: From 0 to 48 hours post dose
Reporting Status: Not Posted

3. Secondary Outcome: Phenolic Acids
Description: Phenolic acids in plasma and urine
Time Frame: 0-48 h post dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: This adverse event occurred during the 1st intervention. The subject did not wish to go on with the study.
Groups:
- Refined Wheat Flour: A treated cereal flour mixed with milk (negative control).
- Esterase Wholegrain Wheat Flour: A cereal flour treated with esterases to release phenolics (positive control for phenolic acids)
Arm/Group | Refined Wheat Flour | Esterase Wholegrain Wheat Flour | Liquid Whole Grain Wheat Flour | Liquid Wholegrain Barley Flour | Wholegrain Wheat Flour | Wholegrain Barley Flour
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refined Wheat Flour (N=14) | Esterase Wholegrain Wheat Flour (N=14) | Liquid Whole Grain Wheat Flour (N=14) | Liquid Wholegrain Barley Flour (N=14) | Wholegrain Wheat Flour (N=14) | Wholegrain Barley Flour (N=14)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The subject complain of nausea in the hour following the product intake and vomitted 8 hours later.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No